CLINICAL TRIAL: NCT04483817
Title: Efficacy of Transcutaneous Versus Percutaneous Posterior Tibial Nerve Stimulation in the Treatment of Overactive Bladder. Randomized Clinical Trial.
Brief Title: Efficacy of Transcutaneous Versus Percutaneous Posterior Tibial Nerve Stimulation in the Overactive Bladder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fisiocore LC,SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 06/2019
Record Dates: First submitted 2020-03-27; First posted 2020-07-23 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Overactive Bladder Syndrome
Keywords: urgency; incontinence; nocturia; frequency
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Intervention Model Description: prospective interventional study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Transcutaneous tibial nerve stimulation (Experimental): The transcutaneous electrostimulation of the posterior tibial nerve (ETNTP) will be applied to group A: place two surface electrodes, one 32 mm in diameter, 5 cm cephalad of the internal malleolus and 1 cm medial posterior of the tibia; and another 50x50 mm electrode in the calcaneous. The flexion of the first toe will indicate the correct placement of the electrodes. Stimulation is performed according to the Stoller method with a stimulator programmed at 20Hz and 200 µs, with a continuous current, 12 sessions, 2 weekly are completed. The intensity of the current will be tolerance by the subject.
  Interventions: Device: Transcutaneous tibial nerve stimulation
- B: Percutaneous tibial nerve stimulation (Active Comparator): The percutaneous electrostimulation of the posterior tibial nerve (EPNTP) will be applied to group B: inserting a 0.25x30mm surgical steel needle at a 60º angle, 5 cm cephalad to the malleolus and 1 cm posterior of the tibia , and a surface electrode of 50x50 mm in the calcaneous. The flexion of the first finger will indicate its correct placement. The stimulation parameters will also follow the Stoller method.
  Interventions: Device: Percutaneous tibial nerve stimulation

INTERVENTIONS:
Device: Transcutaneous tibial nerve stimulation — Apply tibial nerve stimulation with surface electrodes in the treatment of overactive bladder.
  Arms: A: Transcutaneous tibial nerve stimulation
Device: Percutaneous tibial nerve stimulation — Apply tibial nerve stimulation with surface electrodes in the treatment of overactive bladder.
  Arms: B: Percutaneous tibial nerve stimulation

SUMMARY:
The main aim of this study, is compare the effectiveness of transcutaneous posterior tibial nerve stimulation versus percutaneous posterior nerve stimulation in patients with overactive bladder.

DETAILED DESCRIPTION:
Overactive bladder syndrome (OAB) is a set of symptoms characterized by urge, with or without urge incontinence, usually with frequency and nocturia in the absence of urinary infection or other pathologies. OAB affect considerably the quality of life of the subject who suffer.

The first line of treatment is a conservative management as behavioral interventions, followed by pharmacological management as antimuscarinic or antimuscarinic drugs.

Percutaneous tibial nerve stimulation (PTNS) is present as another alternative of treatment. Previous studies have shown the positive effects of PTNS in a reduction on OAB symptoms.

The PTNS was described by Stoller in 1999. It's a electrical stimulation of the tibial nerve, inserting a 34 gauge needle at a 60º angle, 5 cm cephalad to the malleolus and 1 cm posterior of the tibia, to stimulation of the sacral segments S2 and S3, where the spinal centre of bladder is located. The parameters used are 20Hz and 200 µs, 12 sessions, two weekly, 30 min treatment.

The PTNS is a minimal invasive technique, but can be utilized surface electrodes instead of needle to minimize the discomfort of prick.

The main aim of this study, is compare the effectiveness of transcutaneous posterior tibial nerve stimulation versus percutaneous posterior nerve stimulation in patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosis of overactive bladder
* Subjects refractory to treatments antimuscarinic or beta 3-agonist
* Subjects who do not take restricted medication
* Subjects who can cognitively complete the voiding diary and questionnaires
* Subject with symptoms 3 months ago
* Men must be discarded obstruction by benign prostatic hyperplasia

Exclusion Criteria:

* Subjects with stress incontinence
* Subjects with urinary tract infection
* Subjects with neurological disease
* Subjects with pacemakers fitted
* Pregnancy
* Subjects who have disorder sensitive
* A history of pelvic tumors
* Subject who is not able to understand the physiotherapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Urinary frequency | two years
  Urinary episodes per day.
  According to international consensus, it is considered pathological when:
  There are more than 8 episodes of urination per day
Nightime voids | two years
  Urinary episodes per night.
  According to international consensus, it is considered pathological when:
  There is more than 1 episode per night.
Urge episodes | two years
  Urinary urge episodes per day. The degree of urgency is measured through the PPIUS scale (outcome no. 4). A grade 3-4 on the PPIUS scale is considered pathological.
Degree of urge to void | two years
  Measured through the PPIUS (Patient Perception of Intensity of Urgency Scale).
  Scale from 0 to 4, where:
  0 = No urgency;
  1. = Slight urgency;
  2. = Moderate urgency;
  3. = severe urgency;
  4. = urge incontinence.
Voided volume | two years
  Urine 24 hours volume. Voiding volume over 3000cc in 24 hours, is considered pathological.

SECONDARY OUTCOMES:
Overactive Bladder questionnaire Short- Form (OABq-SF) | Two years
  This is a questionnaire that evaluates both the symptoms and the quality of life of the patient:
  * Symptom involvement (6 questions): Score of 6-36
  * Quality of life (13 questions): Score of 13-78
  * 0-100 metric scale. The higher the score, the more severity.
International Consultation on Incontinence Questionnaire (ICIQ-SF) | Two years
  This is a self-administered questionnaire that identifies people with urine incontinence (UI) and also assess the impact on quality of life. ICIQ-SF Score: Adding the scores to questions 1+2+3, a score above zero is considered a diagnosis of UI.
Benefits, satisfaction and willingness to continue to treatment (BSW) | Two years
  The BSD12 questionnaire is a 3 item likert-type questionnaire (benefit, satisfaction and willingness) with an overall score of 0 to 10. Higher scores indicates a better perception of benefit and satisfaction with the treatment, and a greater willingness to continue with it.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Calzado Sanz, Physiotherap, Principal Investigator — Fisiocore LC,SL
Locations (1):
- Laura Calzado Sanz, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wibisono E, Rahardjo HE. Effectiveness of Short Term Percutaneous Tibial Nerve Stimulation for Non-neurogenic Overactive Bladder Syndrome in Adults: A Meta-analysis. Acta Med Indones. 2015 Jul;47(3):188-200. PMID 26586384
- [Result] Yoong W, Ridout AE, Damodaram M, Dadswell R. Neuromodulative treatment with percutaneous tibial nerve stimulation for intractable detrusor instability: outcomes following a shortened 6-week protocol. BJU Int. 2010 Dec;106(11):1673-6. doi: 10.1111/j.1464-410X.2010.09461.x. PMID 20590544
- [Result] Civic D, Black E. Re: Randomized trial of percutaneous tibial nerve stimulation versus sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial: K. M. Peters, D. J. Carrico, R. A. Perez-Marrero, A. U. Khan, L. S. Wooldridge, G. L. Davis and S. A. MacDiarmid J Urol 2010; 183: 1438-1443. J Urol. 2011 Jan;185(1):362; author reply 362-4. doi: 10.1016/j.juro.2010.09.030. Epub 2010 Nov 18. No abstract available. PMID 21092997
- [Result] Sajadi KP, Goldman HB. Percutaneous tibial nerve stimulation and overactive bladder. Curr Urol Rep. 2010 Sep;11(5):293-5. doi: 10.1007/s11934-010-0126-4. No abstract available. PMID 20567947
- [Result] Booth J, Connelly L, Dickson S, Duncan F, Lawrence M. The effectiveness of transcutaneous tibial nerve stimulation (TTNS) for adults with overactive bladder syndrome: A systematic review. Neurourol Urodyn. 2018 Feb;37(2):528-541. doi: 10.1002/nau.23351. Epub 2017 Jul 21. PMID 28731583
- [Result] Burton C, Sajja A, Latthe PM. Effectiveness of percutaneous posterior tibial nerve stimulation for overactive bladder: a systematic review and meta-analysis. Neurourol Urodyn. 2012 Nov;31(8):1206-16. doi: 10.1002/nau.22251. Epub 2012 May 11. PMID 22581511
- See also: Guidelines of urology´s treatments — http://uroweb.org/guidelines/
- See also: Guidelines of AEU (Asociación Española de Urología) — http://www.teknon.es/idcsalud-client/cm/images?idMmedia=444713